CLINICAL TRIAL: NCT06219356
Title: A Phase 1 Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Preliminary Efficacy of GLB-002 in Patients With Relapsed or Refractory Non-Hodgkin Lymphomas (R/R NHL)
Brief Title: A Study of GLB-002 in Patients With Relapsed or Refractory Non-Hodgkin Lymphomas
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Hangzhou GluBio Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GLB-002-01
Record Dates: First submitted 2023-12-22; First posted 2024-01-23 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-06

CONDITIONS: Non-Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Dose Escalation of GLB-002 in Participants with R/R NHL-Phase 1a (Experimental): Part 1a (Dose Escalation) of the study will enroll R/R NHL participants and will evaluate the safety, tolerability, PK, PD and preliminary efficacy of GLB-002 administered orally, and determine the maximum tolerated dose (MTD) and/or recommended expansion doses (RED) in R/R NHL patients who are eligible for dose limiting toxicity (DLT) evaluation.
  Interventions: Drug: GLB-002
- Dose Expansion of GLB-002 in Participants with R/R FL (Grade 1, 2, 3a)-Phase 1b Cohort 1 (Experimental): Part 1b (Dose Expansion) Cohort 1 will confirm tolerability of the selected doses and schedules and evaluate whether efficacy is in a range that warrants further clinical development for R/R Follicular Lymphoma (Grade 1、2、3a).
  Interventions: Drug: GLB-002
- Dose Expansion of GLB-002 in Participants with R/R DLBCL and FL (Grade 3b)-Phase 1b Cohort 2 (Experimental): Confirm tolerability of the selected doses and schedules and evaluate whether efficacy is in a range that warrants further clinical development for R/R Diffuse Large B-cell Lymphoma and R/R Follicular Lymphoma (Grade 3b).
  Interventions: Drug: GLB-002
- Dose Expansion of GLB-002 in Participants with other R/R NHL-Phase 1b Cohort 3 (Experimental): Part 1b (Dose Expansion) Cohort 3 will confirm tolerability of the selected doses and schedules and evaluate whether efficacy is in a range that warrants further clinical development for other R/R NHL, including, but not limited to Mantle-cell Lymphoma (MCL), Marginal Zone Lymphoma (MZL), Small Lymphocytic Lymphoma (SLL) /Chronic Lymphocytic Leukemia (CLL) and Peripheral T-cell Lymphoma (PTCL).
  Interventions: Drug: GLB-002

INTERVENTIONS:
Drug: GLB-002 — Administered orally according to the assigned treatment schedule.
  Other Names: GLB-A062-B

SUMMARY:
Study GLB-002-01 is a first-in-human (FIH), phase 1, open-label, dose escalation and expansion clinical study, the purpose of this study is to evaluate the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD) and preliminary efficacy of GLB-002 monotherapy in participants with relapsed or refractory Non-Hodgkin lymphomas (R/R NHL).

ELIGIBILITY:
Inclusion Criteria:

* Participants must understand and voluntarily sign a written informed consent form (ICF) prior to any study-related assessments/procedures being performed.
* Participants is ≥18 years of age at the time of signing the ICF.
* Participants with histopathologically or immunohistochemically confirmed NHL according to 2016 World Health Organization (WHO) haematolymphoid tumors criteria classification (CLL/SLL diagnosis according to 2018 IWCLL) who have failed standard of care therapy or lack an effective treatment regimen.
* Participants in Phase Ib screening period with measurable lesion, but no measurable nodal lesion limit for participants in Phase Ia.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0,1 or 2.
* Life expectancy > 3 months.
* Good performance of major organs, including hematology, liver and kidney function, and coagulation. etc.
* Participants are willing and able to adhere to the study visit schedule and other protocol requirements.

Exclusion Criteria:

* Receipt of anticancer medications/therapies such as chemotherapy, targeted therapy, immunotherapy, biologic therapy, or herbal agent ≤ 28 days or 5 half-lives, whichever is shorter, prior to the first dose of GLB-002; or chimeric antigen receptor T cell therapy (CAR-T) within 3 months prior to the first dose of GLB-002.
* Currently enrolled in any other investigational drug study or participation within the last 28 days or 5 half-lives, whichever is shorter, prior to the first dose of GLB-002 (exception of participants who participated in only one investigational drug study with overall survival follow-up).
* Participants with unresolved clinically significant toxicities of > Grade 1 AE or not be recovered to baseline value from prior anticancer therapies with exception of alopecia or hyperpigmentation of the skin.
* Participants who are scheduled to receive other anticancer therapies or other investigational drugs during the study period.
* Participants with active acute or chronic graft versus host disease (GVHD) requiring systemic immunosuppressive therapy, or participants requiring treatment with systemic corticosteroids (>10 mg/day prednisone or equivalent) or other immunosuppressive drugs within the last 7 days prior to the first dose of GLB-002 or during the study period.
* Receipt of Autologous Stem Cell Transplantation (ASCT) within the last 3 months, or allogeneic hematopoietic stem cell transplantation (allo-HSCT) within the last 6 months prior to the first dose of GLB-002.
* Participants with known active leukemic involvement in central nervous system (CNS).
* Participants with peripheral neuropathy ≥ Grade 2 (Graded according to CTCAE version 5.0).
* History of, or current active cancer other malignancy for the past 5 years, with the exception of curatively resected cancer in situ, including cervical carcinoma in situ, basal cell carcinoma of the skin, or prostate cancer in situ, etc
* QT interval interval >470 milliseconds (ms) using electrocardiographic (ECG) at Screening.
* Participants has impaired cardiac function or clinically significant cardiac disease at current or within last 6 months.
* Participants with known active infection of hepatitis B virus (HBV) or hepatitis C virus C (HCV).
* Participants with known human immunodeficiency virus (HIV) infection.
* Participants with known life-threatening or clinical significant uncontrolled active systemic infections unrelated to malignant hematologic diseases
* Participants with a condition that may affects the absorption, distribution, metabolism and excretion of GLB-002.
* Medications or supplements that are known to be strong and moderate inhibitors or inducers of cytochrome P-450 isozyme (CYP)3A4/5 and/or P-glycoprotein (P-gp) within 7 days or 5 half-lives prior to the first dose of GLB-002, whichever is shorter.
* Participants who have undergone major surgery within 28 days prior to the first dose of the GLB-002.
* Pregnant or lactating women.
* Participants who have cognitive impairment due to any psychiatric or neurological condition, including epilepsy and dementia, may limit their understanding, performance, and study compliance with the ICF.
* Participants,in the opinion of the Investigator, who are unsuitable to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2024-01-11 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting Toxicity (DLT) | Up to 35 days after first dose of study treatment in Phase 1a
  DLT is defined as the treatment emergent adverse events (TEAEs) meeting protocol specified DLT criteria and occurring within the DLT assessment period, except those that are clearly and incontrovertibly due to extraneous causes including disease progression, pre-existing medical condition that has not worsened from baseline, or other causes that are clearly not due to study drug.
Maximum Tolerated Dose (MTD) | Up to 2 years (each cycle is 28 days)
  MTD is defined as the highest dose level at which no more than 1 of 6 DLT-evaluable participants experienced a DLT.
Recommended Expansion Doses (RED) | Up to 2 years (each cycle is 28 days)
  RED will be decided by safety review committee (SRC) considering the data including safety, tolerability, PK, PD, and preliminary efficacy of GLB-002 in dose escalation. RED will be the dose level below MTD.
Incidence, Relatedness, Seriousness and Severity of Adverse Events (AEs) | Up to 2 years
  AE is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. AE will be graded according to the National Cancer Institute Common Terminology Criteria for AE (NCI CTCAE) version 5.0.
Recommended Phase 2 Dose (RP2D) | Up to 2 years
  RP2D based on the totality of data across dosing cohorts in the dose escalation and expansion phases of the study including PK, PD, safety and efficacy outcomes.
Objective Response Rate (ORR) | Up to 2 years
  ORR is defined as the percent of participants whose best overall response is complete response (CR) or partial response (PR). CR and PR will be assessed by 2014 Lugano for NHL and/or 2018 International Working Group Criteria for Chronic Lymphocyte Leukemia (2018 IWCLL).
Time to Response (TTR) | Up to 2 years
  For participants with objective response, TTR was defined as the time of participants from the first treatment administration to the first incidence of a confirmed CR or PR was reported. CR and PR will be assessed by 2014 Lugano for NHL and/or 2018 IWCLL.
Duration of Remission or Response (DOR) | Up to 2 years
  For participants with objective response, DOR is measured from the time of any of CR or PR are first met (whichever is first recorded) until the first date at which progressive disease or death from any cause is objectively documented assessment. CR and PR will be assessed by 2014 Lugano for NHL and/or 2018 IWCLL.
Progression-free Survival (PFS) | Up to 2 years
  PFS is defined as the time from the first dose of GLB-002 to the first occurrence of progressive disease (PD) or death from any cause. PD will be assessed by 2014 Lugano for NHL and/or 2018 IWCLL.
Overall Survival (OS) | Up to 2 years
  OS is defined as the time from the first dose of GLB-002 to death due to any cause.

SECONDARY OUTCOMES:
GLB-002 and GLB-A062-A (R-enantiomers of GLB-002) Pharmacokinetics after Single Administration-AUC0-last | Up to 48 hours after single administration
  Area under the concentration-time curve from zero to the last measurable concentration
GLB-002 and GLB-A062-A Pharmacokinetics after Single Administration-AUC0-24 | Up to 48 hours after single administration
  Area under the concentration-time curve from 0 to 24 hours
GLB-002 and GLB-A062-A Pharmacokinetics after Single Administration-AUC0-inf | Up to 48 hours after single administration
  Area under the concentration-time curve from 0 to infinity
GLB-002 and GLB-A062-A Pharmacokinetics after Single Administration-Cmax | Up to 48 hours after single administration
  Maximum plasma concentration
GLB-002 and GLB-A062-A Pharmacokinetics after Single Administration-Tmax | Up to 48 hours after single administration
  The time to reach maximum concentration
GLB-002 and GLB-A062-A Pharmacokinetics after Single Administration-T1/2 | Up to 48 hours after single administration
  Terminal half-life
GLB-002 and GLB-A062-A Pharmacokinetics after Single Administration-Vz/F | Up to 48 hours after single administration
  Apparent volume of distribution
GLB-002 and GLB-A062-A Pharmacokinetics after Single Administration-CL/F | Up to 48 hours after single administration
  Apparent total clearance of the drug from plasma after oral administration
GLB-002 and GLB-A062-A Pharmacokinetics after Single Administration-λz | Up to 48 hours after single administration
  Terminal rate constant
GLB-002 and GLB-A062-A Pharmacokinetics after Multiple Administration-Tmax,SS | Up to 2 years
  Time of maximum concentration at steady state
GLB-002 and GLB-A062-A Pharmacokinetics after Multiple Administration-Cav,SS | Up to 2 years
  Average plasma concentration at steady state
GLB-002 and GLB-A062-A Pharmacokinetics after Multiple Administration-Cmax,SS | Up to 2 years
  Maximum plasma concentration at steady state
GLB-002 and GLB-A062-A Pharmacokinetics after Multiple Administration-Cmin,SS | Up to 2 years
  Minimum plasma concentration at steady state
GLB-002 and GLB-A062-A Pharmacokinetics after Multiple Administration-AUC0-tau | Up to 2 years
  Area under the concentration-time curve during the dosing interval
GLB-002 and GLB-A062-A Pharmacokinetics after Multiple Administration-λz | Up to 2 years
  Terminal rate constant
GLB-002 and GLB-A062-A Pharmacokinetics after Multiple Administration-Vz/F | Up to 2 years
  Apparent volume of distribution
GLB-002 and GLB-A062-A Pharmacokinetics after Multiple Administration-CLSS/F | Up to 2 years
  Apparent clearance at steady state
GLB-002 and GLB-A062-A Pharmacokinetics after Multiple Administration-T1/2 | Up to 2 years
  Terminal half-life
GLB-002 and GLB-A062-A Pharmacokinetics after Multiple Administration-Rac [AUC] | Up to 2 years
  Accumulation index in area under the concentration-time curve
GLB-002 and GLB-A062-A Pharmacokinetics after Multiple Administration-Rac [Cmax] | Up to 2 years
  Accumulation index in maximum plasma concentration
GLB-002 and GLB-A062-A Pharmacokinetics after Multiple Administration-DF | Up to 2 years
  Degree of fluctuation index

CONTACTS AND LOCATIONS:
Overall Officials: Gang Lu, Ph.D., Study Director — Hangzhou GluBio Pharmaceutical Co., Ltd.
Locations (13):
- China (13):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - Jiangxi Cancer Hospital, Nanchang, Jiangxi
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Shanxi Cancer hospital, Taiyuan, Shanxi
  - Tianjing Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality
  - The First Affilicated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang